CLINICAL TRIAL: NCT03580980
Title: Evaluation of Multimodal Preemptive Analgesia in Major Pediatric Abdominal Cancer Surgeries
Brief Title: Multimodal Analgesia in Major Abdominal Pediatric Cancer Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ehab Hanafy Shaker, Clinical professor of Anesthesia ,Critical care and Pain medicine, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Ehab-Hossam.multi
Record Dates: First submitted 2018-06-23; First posted 2018-07-10 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Pediatric Cancer; Pain, Postoperative
MeSH Terms: conditions — Neoplasms; Pain, Postoperative | interventions — Acetaminophen; Ketamine; Combined Modality Therapy; Injections, Epidural; Morphine; Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Drug: Morphine (Active Comparator): Morphine Group C (n=30) was the control group who received IV morphine in a dose of 0.1 mg/kg after induction of anesthesia
  Interventions: Drug: Morphine
- Procedure/surgery:Caudal levobupivacaine (Active Comparator): In Caudal Group (n=30), patients were placed in the lateral position and received caudal epidural block after induction of anesthesia with levobupivacaine 0.125% , 1.1 ml/kg and morphine 0.02 mg/kg with maximum 20ml.
  Interventions: Procedure: Caudal levobupivacaine
- Drug: Paracetamol and ketamine (Active Comparator): The patients of Multimodal Group (n=30) received paracetamol infusion 10 mg/kg over 10 minutes and ketamine 0.5 mg/kg IV bolus followed by ketorolac 1 mg/kg infusion over 10 minutes.
  Interventions: Drug: Paracetamol and ketamine

INTERVENTIONS:
Drug: Paracetamol and ketamine — intravenous paracetamol and ketamine followed by ketorolac
  Other Names: Multimodal
  Arms: Drug: Paracetamol and ketamine
Procedure: Caudal levobupivacaine — an epidural injection of morphine and levobupivacaine through the caudal space
  Other Names: Epidural
  Arms: Procedure/surgery:Caudal levobupivacaine
Drug: Morphine — patient controlled analgesia by morphine
  Other Names: Patient controlled analgesia
  Arms: Drug: Morphine

SUMMARY:
Surgical trauma initiates multiple physiological mechanisms that cause postoperative pain. Postoperative pain has nociceptive, inflammatory, and neuropathic components.Inadequate relief of postoperative pain leads to significant morbidity, delayed recovery, and mortality.Adverse reactions of medications used for postoperative pain management, particularly opioids, are common including pruritus and nausea and vomiting.Preemptive analgesia is defined as analgesic treatment that starts before surgical incision to prevent central sensitization caused by incisional and inflammatory injuries.Therefore, in this pilot study, the investigators are trying to evaluate safety and efficacy of preemptive multimodal analgesia compared with preemptive caudal analgesia and PCA morphine in pediatric cancer patient undergoing major abdominal surgery.

DETAILED DESCRIPTION:
Surgical trauma initiates multiple physiological mechanisms that cause postoperative pain. Postoperative pain has nociceptive, inflammatory, and neuropathic components.Inadequate relief of postoperative pain leads to significant morbidity, delayed recovery, and mortality.Despite the development of new drugs and analgesic techniques, up to 40% of hospitalized children - especially surgical patients - experiences moderate to severe pain. Adverse reactions of medications used for postoperative pain management, particularly opioids, are common including pruritus and nausea and vomiting.The incidence of opioid-related respiratory depression was reported to range from 0.11 to 0.41%.Regional anesthesia was suggested as an alternative to opioid-based analgesia in pediatric patients. Caudal epidural analgesia is a relatively safe and simple technique for postoperative pain management in children.However, there is a potential for adverse effects related to the technique of catheter placement or systemic toxicity of the local anesthetic.

Preemptive analgesia is defined as analgesic treatment that starts before surgical incision to prevent central sensitization caused by incisional and inflammatory injuries.However, studies in animal models of incisional pain demonstrated that single analgesic treatment before the incision does not reduce postoperative pain. Once nociceptive afferent block subsides, the wound reinitiates central sensitization. Also, clinical trials reported similar results.Multimodal analgesia uses a combination of delivery routes administered at variable time points to optimize outcomes in the treatment of acute pain.

Therefore, in this pilot study, the investigators are trying to evaluate safety and efficacy of preemptive multimodal analgesia compared with preemptive caudal analgesia and PCA morphine in pediatric cancer patient undergoing major abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* were ASA I or II patients.
* Aged between 5 and 12 years.
* Both sexes.
* Scheduled for major abdominal surgery with a midline incision.

Exclusion Criteria:

* included history of mental retardation or delayed development that may interfere with pain intensity assessment,
* Known or suspected allergy to any administered drugs.
* Active renal (creatinine clearance <50).
* Hepatic (liver enzymes more than 10 folds).
* Respiratory (SPO2 <92% on room air).
* Cardiac disease (ejection fraction < 50%).

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours
  Total morphine consumption during the postoperative 24 hours

SECONDARY OUTCOMES:
Changes in VAS score for pain | Baseline and 6,12,18 and 24 hours
  it is a scoring system from 0 to 100 where 0 means no pain while 100 represents maximum pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ehab H Shaker, MD, Principal Investigator — National Cancer Institute- Cairo University
Locations (1):
- Department of Anesthesia and Pain medicine.National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
after submission of the study it will be available for all researchers through the publication